CLINICAL TRIAL: NCT06264726
Title: CommunityRx-Cardiovascular Disease: Implementation of the HealtheRx to Reduce Health Inequity in Rural Eastern North Carolina
Brief Title: CommunityRx-Cardiovascular Disease
Acronym: CRx-CVD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-0254; R01HL150909 (NIH)
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Self Efficacy
Keywords: cardiovascular disease; social determinants of health; rural health; health related social needs; self efficacy
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): This group will receive the intervention
  Interventions: Other: HealtheRx

INTERVENTIONS:
Other: HealtheRx — CRx-CVD intervention provides participants with a HealtheRx, a tool developed by researchers with personalized listings of community resources with information about housing, food assistance, utility support, transportation and crisis support for patients. A HealtheRx may can be given directly, texted or emailed to patients and caregivers. All patients enrolled in this group will receive the HealtheRx either via text and/or email based on participant preference. Participants will receive contact information for a Community Resource Navigator who can provide support with using the HealtheRx, provide additional resources upon request, and answer any questions the participant may have. Participants will also receive a 2 reminder text messages over 2 months following their initial receipt of the HealtheRx. The SMS messages offer reminders about the HealtheRx and ongoing community resource navigation support.

SUMMARY:
The goal of this single arm pre-test post-test design study is to test the impact of providing patients with information about community-based resources to address health-related social needs and cardiometabolic health in rural African American patients. The main question it aims to answer is:

• What is the effectiveness of community resource information on patient self-efficacy to use community resources?

Participants will be given:

* A personalized "HealtheRx" resource with information about community resources related to food, housing, utility support, transportation, and crisis support. The HealtheRx is personalized for patients based on their age and zip code.
* Access to a community resource navigator for support with using the HealtheRx upon request
* 2 text messages with reminders about the HealtheRx and access to the community resource navigator

ELIGIBILITY:
Inclusion Criteria:

* patient
* African American
* age 2 or older
* Have at least one cardiometabolic condition:

  * Overweight (BMI greater than or equal to 25 kg/m^2);
  * Obesity (BMI greater than or equal to 30 kg/m^2);
  * ICD-9 or 10 diagnostic code for overweight or obesity
  * Adult prehypertension (SBP 120 to 129 and DBP greater than 80 mmHg);
  * Adult hypertension (SBP greater than or equal to130 or DBP = 80 mmHg);
  * Pediatric Prehypertension (SBP or DBP greater than or equal to 90th but <95th percentile)
  * Pediatric Hypertension (SBP or DBP greater than or equal to 95th percentile);
  * ICD-9 or 10 diagnostic code for hypertension
  * Adult and Pediatric Prediabetes (Fasting glucose 100-125 mg/dL or OGTT 140-199 mg/dL)
  * Adult and Pediatric Diabetes (FPG greater than or equal to126 mg/dL (7.0 mmol/L) or OGTT greater than or equal to 200 mg/dL (11.1mmol/L) or HgbA1C greater than or equal to 6.5);
  * ICD-9 or 10 diagnostic code for diabetes, pre-diabetes or elevated glucose, or gestational diabetes;
  * Adult and Pediatric Total cholesterol (>200mg/dL; LDL >130mg/dL; HDL < 35 mg/dL; TG greater than or equal to150mg/dL);
  * ICD-9 or 10 diagnostic code for hyperlipidemia

Exclusion Criteria:

* Unable to read, speak or understand English
* Unable to receive text message or email communications
* Living in the same household as someone already enrolled in the CRx-CVD study
* Adults with limited life expectancy (e.g., advanced cancer, end stage liver disease, hospice)
* Adults receiving treatment for cancer
* Adults living in skilled nursing facilities
* Dementia/other significant cognitive impairment

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in participant self-efficacy for finding community resources | Baseline, up to 6 months
  Change in self-efficacy for finding community resources is measured using one item constructed from Bandura's Self-Efficacy Scale which asks, "How confident are you in your ability to find resources in your community that help you manage your health?" Responses will be assessed on a 5-point Likert scale ranging from 1= "not at all confident" to 5= "completely confident." Lower scores indicate lower levels of confidence, and higher scores indicate higher levels of confidence. We will report counts with percentages pre- and post-intervention.

SECONDARY OUTCOMES:
Change in participant knowledge of community resources | Baseline, up to 6 months
  Change in participant knowledge of community resources is measured using 10 self-reported survey items adapted and tested in prior CommunityRx studies asking, "For each place that I list, please tell me if you know of places like this in your community: [insert community resource]." The following responses will be assessed: Yes, no, don't know, refused. We will report counts and percentages for knowledge of 0, 1, 2, 3 or 4 or more resource types pre- and post-intervention.
Change in participant utilization of community resources | Baseline, up to 6 months
  Change in participant utilization of community resources is measured using 10 self-reported survey items adapted and tested in prior CommunityRx studies asking participants "Have you received services from places like this for you or your household in the last 6 months?" The following responses will be assessed: Yes, no, don't know, refused. We will report counts and percentages for utilization of 0, 1, 2, 3 or 4 or more resource types pre- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Dave, MBBS, DrPH, Principal Investigator — Unviersity of North Carolina at Chapel Hill
Locations (2):
- United States (2):
  - OIC Family Medical Center - Fairview, Rocky Mount, North Carolina
  - OIC Family Medical Center - Happy Hill, Rocky Mount, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC